CLINICAL TRIAL: NCT03596515
Title: Occupational Therapy With Ayres Sensory Integration Approach for School-age Children - a Randomized Controlled Trial
Brief Title: Occupational Therapy With Ayres Sensory Integration Approach for School-age Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Phoebe Chan, Occupational Therapist I, Occupational Therapy Department, Principal Investigator, Hong Kong Children's Hospital, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KC/KE-13-0135/FR-3
Record Dates: First submitted 2018-07-02; First posted 2018-07-24 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Children, Only

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Received sensory integration therapy (Experimental): Participants in the experimental group received 16 sessions (45 minutes each) of individualized Ayres Sensory Integration intervention.
  Interventions: Other: Sensory Integration
- Waitlist control group (No Intervention): Participants in the control group received Ayres Sensory Integration according to the usual clinical scheduling. It is after the post- assessment outcome at the same time of the experimental group.

INTERVENTIONS:
Other: Sensory Integration — Sensory Integration (SI) is a theory and framework conceptualized by Dr. Jean Ayres, a highly experienced occupational therapist, with its main objective as enhancing the brain's capacity to perceive and organize sensory information to produce a more normal, adaptive response; thus, to provide the foundation for mastering academic tasks.
  Other Names: Ayres Sensory Integration Approach
  Arms: Received sensory integration therapy

SUMMARY:
Introduction:

Sensory Integration (SI) is a theory and framework conceptualized by Dr. Jean Ayres, a highly experienced occupational therapist, with its main objective as enhancing the brain's capacity to perceive and organize sensory information to produce a more normal, adaptive response; thus, to provide the foundation for mastering academic tasks (Case-Smith and O'Brien, 2010).

Objectives:

The aim of the study is to investigate the effectiveness of ASI interventions for school-aged children with sensory modulation and sensory processing deficits.

Methodology:

A cross-clustered single-blinded randomized controlled trial was conducted in 5 occupational therapy outpatient department within Hospital Authority, to assess the difference in clinical outcomes between subjects in experimental group (received ASI) and control group (on usual waitlist for treatment). Participants in experimental group (EG) would receive 16 sessions (45 minutes each) of individualized ASI. The sessions were scheduled on weekly basis and would be completed within five months once treatment was initiated. Post-assessment outcomes would be measured at this time-point. Post-assessment outcomes would also be measured for subjects in control group (CG) at the same time-point. ASI would then be initiated for participants in CG according to usual clinical scheduling.

ELIGIBILITY:
Inclusion Criteria:

* aged between six and 12 years old, and attending mainstream primary school
* identified as having problems with sensory modulation and/or sensory processing, according to the Sensory Integration and Praxis Test (SIPT) and the Chinese Sensory Profile completed by their main caregivers for pre-treatment evaluation (definite differences on at least three out of seven of the factor summary or section summary)
* absence of serious emotional or behavioral disturbance
* intelligence quotient no lower than limited (scores range from limited to average or above average).

Exclusion Criteria:

* any neurological problem, such as cerebral palsy
* a history of visual and/or auditory defects or physical problems

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change on the Goal attainment scaling. Changes in functional goals were measured using goal attainment scaling in collaboration with parents and caregivers. | Pre and post of the treatment intervention, an average of 5 months
  Goal attainment scaling (GAS) is the full name of this scale. It is an individualized, criterion-referenced measures of changes. In involves defining a set of unique goals for a client, and then specifying a range of outcomes, which reflect concrete activities. It is a goal-setting process determining intervention outcomes expressly relevant to individuals and their families. It can show functional and meaningful outcomes that are often challenging to assess using standardized measures. It is a 5-point rating scale ranging from -2 to +2 (-2 is the least favorable treatment outcome, 0 is the predicted expected level of performance, and +2 is the most favorable treatment outcome). In this study, three individualized goals were developed for each participant by occupational therapists in conjunction with the parents or caregivers. The occupational therapists transferred the score of each child in each goal in the pre- and post-assessments according to parents' ratings.
Change on the Sensory Integration and Praxis Test scores | Pre and post of the treatment intervention, an average of 5 months
  Sensory Integration and Praxis Test (SIPT) is the full name of this scale. This is a standardized test for assessing the sensory integration and praxis of children between the ages of four years and eight years, eleven months. This study used six subtests of the SIPT - standing and walking balance, postural praxis, post-rotary nystagmus, motor accuracy, sequencing praxis, and graphesthesia - based on expert opinions. SIPT offers is computer scoring and interpretation. Therapists simply record the child's performance and enter into the software. The software will generates the S.D. scores and percentile scores. Average SD scores are usually considered to fall between -1 to +1. Scores below -2 generally indicate definite problems, while scores between -2 and -1 are indicative of possible problems.
Change on the Chinese Sensory Profile | Pre and post of the treatment intervention, an average of 5 months
  Chinese Sensory Profile is the full name of this scale.This is a judgment-based questionnaire answered on a 5-point Likert scale. It is regarded as a standardized assessment for screening the sensory processing abilities of children between the ages of three and 12 years. Score each response according to the following criteria:1. Always = 1 point; 2. Frequently = 2 points; 3. Occassionally = 3 points; 4. Seldom = 4 points; 5. Never = 5 points.To determine the section raw score total, add the item scores for each section and transfer the total to the section summary table. Plot the child's section raw score totals in the classification column corresponding to the raw score total for each section.Cut scores were determined for each section in the following manner: 1. Typical performance includes scores at or above 1 S.D. below the mean; 2. Probable difference is includes scores at or above 2 S.D. below the mean; 3. Definite difference is includes scores below 2 S.D. below the mean.

REFERENCES:
- [Background] Miller LJ, Coll JR, Schoen SA. A randomized controlled pilot study of the effectiveness of occupational therapy for children with sensory modulation disorder. Am J Occup Ther. 2007 Mar-Apr;61(2):228-38. doi: 10.5014/ajot.61.2.228. PMID 17436845
- [Background] Roberts JE, King-Thomas L, Boccia ML. Behavioral indexes of the efficacy of sensory integration therapy. Am J Occup Ther. 2007 Sep-Oct;61(5):555-62. doi: 10.5014/ajot.61.5.555. PMID 17944293
- [Background] May-Benson TA, Koomar JA. Systematic review of the research evidence examining the effectiveness of interventions using a sensory integrative approach for children. Am J Occup Ther. 2010 May-Jun;64(3):403-14. doi: 10.5014/ajot.2010.09071. PMID 20608272
- [Background] Case-Smith J, Weaver LL, Fristad MA. A systematic review of sensory processing interventions for children with autism spectrum disorders. Autism. 2015 Feb;19(2):133-48. doi: 10.1177/1362361313517762. Epub 2014 Jan 29. PMID 24477447
- [Result] Candler C. Sensory integration and therapeutic riding at summer camp: occupational performance outcomes. Phys Occup Ther Pediatr. 2003;23(3):51-64. PMID 14664311